CLINICAL TRIAL: NCT02642679
Title: Evaluation of Opticell Ag (Chitosan Based Dressing) on Split-Thickness Skin Graft (STSG) Donor Sites in Adult Subjects
Brief Title: Evaluation of Opticell Ag on Split-Thickness Skin Graft Donor Sites in Adult Subjects
Acronym: STSG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Medline Industries (Industry)
Responsible Party: Principal Investigator, Indranil Sinha, Assistant Professor of Surgery, Harvard Medical School, Division of Plastic Surgery, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015P001975
Record Dates: First submitted 2015-12-22; First posted 2015-12-30 (Estimated); Results first posted 2017-12-08 (Actual); Last update posted 2017-12-08 (Actual); Status verified 2017-11

CONDITIONS: Split-thickness Skin Graft Donor Sites
Keywords: Split-thickness skin graft, donor site, chitosan, dressing

STUDY DESIGN:
Intervention Model Description: Opticell Ag dressing applied to STSG donor site
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Opticell Ag (Experimental): Opticell Ag covered with a transparent occlusive dressing (Tegaderm) with evenly distributed perforations which permit a controlled leakage into a layer of cotton gauze pads placed directly over the Opticell Ag and occlusive dressing combination.
  Interventions: Device: Opticell Ag

INTERVENTIONS:
Device: Opticell Ag — Opticell Ag+ applied to STSG donor site
  Other Names: Opticell Ag+; Opticell Ag Plus Gelling Fiber with Silver

SUMMARY:
The purpose of this single center, prospective case series is to evaluate the effective management of split-thickness skin graft donor site wounds using Opticell Ag (Chitosan-based dressing).

ELIGIBILITY:
Inclusion Criteria:

* Inpatient status at study site
* Subject must be receiving a split-thickness skin graft (STSG)
* Wounds must not exceed 10% total body surface area (TBSA)
* Any donor site
* Ability to comply with necessary wound care/follow up

Exclusion Criteria:

* Subject is pregnant
* Subject has been diagnosed with Diabetes
* Subject is a smoker
* Subject takes steroids
* Subject is sensitive and/or allergic to shellfish and/or silver
* Wounds that exceed 10% total body surface area (TBSA)
* Inability to comply with necessary wound care/follow up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Indranil Sinha, MD, Principal Investigator — Brigham and Women's Hospital

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients scheduled to undergo split-thickness skin graft harvesting in the Divisions of Burn and Plastic Surgery at the Brigham and Women's Hospital during the period of time from January to December 2016 were identified as possible study candidates.
Pre-assignment Details: Enrolled participants were excluded from the study prior to experimental dressing application if they were found unable to comply with necessary wound care/follow up, or if their surgeon requested they no longer be enrolled.
Period: Overall Study
Arm/Group | Opticell Ag
Started | 19
Completed (Three patients were withdrawn for personal reasons, and surgeon request.) | 16
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: Subjects undergoing split-thickness autografting by the burn or plastic surgery services at the Brigham and Women's Hospital.
Arm/Group | Opticell Ag
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 15
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19
Allergies to chitosan/shellfish [Count of Participants; unit: Participants] | 0
Reason for split-thickness skin graft [Count of Participants; unit: Participants]
  Burn | 16
  Soft tissue defect | 3
Donor site area [Mean (Full Range); unit: square centimeters] | 196.9 [17.5 to 440]
Dermatome setting [Mean (Full Range); unit: inches] | 0.0122 [0.011 to 0.014]

OUTCOME MEASURES:

1. Primary Outcome: Pain
Description: Pain reported by Subject using a visual analog scale (VAS). This scale measures an unidimensional measure of pain intensity by means of a continuous scale comprised of a horizontal line, 10 centimeters (100 mm) in length. The left side of the scale signifies no pain (score of 0), and the right side the other extreme, worst pain imaginable (score of 10). Patients are asked to place a line perpendicular to the VAS scale at the point that represents their pain intensity.
Time Frame: Assessed up to 14 days of use
Population: Pain was evaluated on postoperative day 1, before the dressing was changed on days 5-7, and before and after dressing removal on days 10-14 using the Visual Analog Scale (VAS). The patient was asked to mark his/her pain level on the line between the two endpoints.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Opticell Ag
Number analyzed (Participants) | 16
units on a scale
  Mean Day 1 | 4.2 (3.2)
  Mean Day 5-7 | 2.5 (2.2)
  Mean Day 10-14 | 1.1 (1)
Statistical Analysis 1: Comparison: Opticell Ag; Test type: Other — We set alpha=0.05/3=0.17 to account for multiple outcomes for sample size and power calculations. With 10 patients in each group, we had 95% power to detect an improvement of 2 points in VAS score assuming a common standard deviation of 1 point with a two sided two sample t-test each at alpha=0.17 level; A student t-test was used for correlated samples to determine if there were significant differences in pain. Microsoft Excel 2010 (Microsoft Corp., Redmond, WA) was used for statistical analysis. Data that were considered normally distributed are reported as the mean ± standard deviation (SD) and percentage. P-values <0.05 were considered significant

2. Primary Outcome: Wound Healing Rate (Re-epithelialization)
Description: The extent of re-epithelialization was evaluated by the surgeon and a blinded expert using photographs taken on days 10-14 and at 1 month postoperatively.
Time Frame: Assessed up to 1 month postoperatively.
Measure: Mean (Standard Deviation); unit: percent (%)
Arm/Group | Opticell Ag
Number analyzed (Participants) | 16
percent (%)
  Day 10-14 | 92.3 (8.9)
  1 month | 99.5 (1)
Statistical Analysis 1: Comparison: Opticell Ag; Test type: Other — We set alpha=0.05/3=0.17 to account for multiple outcomes for sample size and power calculations. With 10 patients in each group, we will have 80% power to detect an improvement in re-epithelialization from 14.6 days to 10 days assuming a common standard deviation of 2.9 days; A student t-test was used for correlated samples to determine if there were significant differences in healing rate. Microsoft Excel 2010 (Microsoft Corp., Redmond, WA) was used for statistical analysis. Data that were considered normally distributed are reported as the mean ± standard deviation (SD) and percentage. P-values <0.05 were considered significant

3. Secondary Outcome: Wound Healing Quality
Description: Assessed using the Vancouver scar scale (VSS) 1-month post-operatively. The VSS is a widely used scale in clinical practice to document change in scar appearance. The scale scores four parameters: pigmentation, vascularity, pliability, and height for a total of 13 points. Normal appearance in each of the parameters garners a score of 0 and scores get higher (2-3) as an increase in parameters is observed. The lower the score, the better the outcome.
Time Frame: Assessed up to 1 month of use
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Opticell Ag
Number analyzed (Participants) | 16
units on a scale | 3 (1.4)
Statistical Analysis 1: Comparison: Opticell Ag; Test type: Other — We set alpha=0.05/3=0.17 to account for multiple outcomes for sample size and power calculations. With 10 patients in each group, we will have 95% power to detect an improvement of 2 points in VSS score assuming a common standard deviation of 1 point; A student t-test was used for correlated samples to determine if there were significant differences in healing quality. Microsoft Excel 2010 (Microsoft Corp., Redmond, WA) was used for statistical analysis. Data that were considered normally distributed are reported as the mean ± standard deviation (SD) and percentage. P-values <0.05 were considered significant

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from January to December 2016.
Description: Although no adverse effects were expected in this study, any occurrence was reported to the Brigham and Women's Hospital/Harvard Medical School IRB within 5 days while following the Partners Human Research Committee Guidelines for Adverse Event Reporting.
Arm/Group | Opticell Ag
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 0/19

LIMITATIONS AND CAVEATS:
This pilot study is not a randomized, control study and is limited by the absence of a small sample size and direct comparison group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No